CLINICAL TRIAL: NCT01772758
Title: Influence of Cystic Fibrosis on Vascular Endothelial Function at Rest and During Exercise
Brief Title: Cystic Fibrosis and Endothelial Function: At Rest and During Exercise
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Ryan Harris, Principal Investigator, Augusta University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CFD Study
Record Dates: First submitted 2012-10-16; First posted 2013-01-21 (Estimated); Results first posted 2018-01-10 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Cystic Fibrosis
Keywords: CF, cystic fibrosis, exercise
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity | interventions — sapropterin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Protocol 1: AOC (Experimental): measurements at baseline and 2 hours following the antioxidant cocktail that is comprised of over the counter vitamins (vitamin C 1000mg, vitamin E 600 IU, and alpha lipoic acid 600 mg) that will be given in two doses, 30 minutes apart.
  Interventions: Dietary Supplement: Antioxidant Cocktail
- Protocol 2: BH4 (5mg) (Experimental): measurements at baseline and 3 hours following the single dose of 5mg/kg Kuvan® or sapropterin dihydrochloride which is a synthetic preparation of the dihydrochloride salt of naturally occurring tetrahydrobiopterin (BH4).BH4 has been shown in past studies to increase NO bioavailability.
  Interventions: Drug: BH4 5mg
- Protocol 2: BH4 (20mg) (Experimental): measurements at baseline and 3 hours following the single dose of 20mg/kg Kuvan® or sapropterin dihydrochloride which is a synthetic preparation of the dihydrochloride salt of naturally occurring tetrahydrobiopterin (BH4).BH4 has been shown in past studies to increase NO bioavailability.
  Interventions: Drug: BH4 20mg
- Healthy Controls (No Intervention): baseline measurements were done with no intervention

INTERVENTIONS:
Drug: BH4 5mg — Kuvan® or sapropterin dihydrochloride is a synthetic preparation of the dihydrochloride salt of naturally occurring tetrahydrobiopterin (BH4). Subjects received an oral dose of 5 mg/kg of Kuvan® (Biomarin Pharmaceuticals Inc.)
  Other Names: Tetrahydrobiopterin; Kuvan
  Arms: Protocol 2: BH4 (5mg)
Drug: BH4 20mg — Kuvan® or sapropterin dihydrochloride is a synthetic preparation of the dihydrochloride salt of naturally occurring tetrahydrobiopterin (BH4). Subjects received an oral dose of 20 mg/kg of Kuvan® (Biomarin Pharmaceuticals Inc.)
  Other Names: Tetrahydrobiopterin; Kuvan
  Arms: Protocol 2: BH4 (20mg)
Dietary Supplement: Antioxidant Cocktail — Vitamin C (1000 mg) , Vitamin E (600 IU) , and alpha-lipoic acid (600 mg). all BID
  Arms: Protocol 1: AOC

SUMMARY:
Perhaps one of the most disturbing aspects of Cystic Fibrosis (CF) is the associated premature death. Oxidative stress has been observed in patients with CF and exercise intolerance has been shown to predict mortality in patients with CF, regardless of how healthy their lungs are. A critical barrier to improving the quality of life and longevity in patients with CF is our lack of knowledge regarding the different reasons why patients with CF cannot exercise to the level of their peers. We have collected preliminary data to support our central hypothesis that oxidative stress contributes to the impairment in blood vessel function at rest and during exercise which ultimately oxygen transport and delivery resulting in exercise intolerance. Exercise is therapeutic medicine for patients with CF and this investigation represents a major breakthrough in the approach to begin understanding the physiological mechanisms which contribute to exercise intolerance in these patients.

DETAILED DESCRIPTION:
The overall goals of this proposal are to provide mechanistic evidence that oxidative stress contributes to 1) endothelial dysfunction and 2) exercise intolerance in patients with CF. This study consists of two separate sub-studies, or protocols. Protocol 1: AOC tested the effect of an antioxidant cocktail (AOC) on endothelial function at rest and during exercise in CF patients. Protocol 2: BH4 tested the effect of tetrahydrobiopterin (BH4) on endothelial function at rest and during exercise in CF patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF and healthy controls
* Men and women (> 18 yrs. old)
* Boys and girls (7 -17 yrs. old)
* FEV1 percent predicted > 30%
* Resting oxygen saturation (room air) >90%
* Patients with or without CFRD
* Traditional CF-treatment medications
* Ability to perform reliable/reproducible PFTs
* Clinically stable for 2 weeks (no exacerbations or need for antibiotic treatment within 2 weeks of testing or major change in medical status)

Exclusion Criteria:

* Children 6 yrs. old and younger
* FEV1 percent predicted < 30%
* Resting oxygen saturation (room air) < 90%
* Clinical diagnosis of heart disease
* Pulmonary artery hypertension
* Febrile illness within two weeks of visit
* Current smokers
* Currently pregnant or nursing
* Individuals on vaso-active medications (i.e. nitrates, beta blockers, ACE inhibitors, etc.)
* Inability to swallow pills
* Patients with B. Cepacia (only ~3% of our CF center patient population)

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-08; Primary Completion 2016-06-21 (Actual); Study Completion 2016-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Harris, PhD, CES, Principal Investigator — Augusta University
Locations (1):
- Georgia Prevention Institute/ Laboratory of Integrative and Exercise Physiology, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Laboratory of Integrative and Exercise Physiology Website — http://facebook.com/harrislab

RESULTS

PARTICIPANT FLOW:
Groups:
- Protocol 1: AOC: measurements at baseline and 2 hours following the antioxidant cocktail that is comprised of over the counter vitamins (vitamin C 1000mg, vitamin E 600 IU, and alpha lipoic acid 600 mg) that will be given in two doses, 30 minutes apart.
  Vitamin C, 1000mg: Vitamin C (1000 mg) , Vitamin E (600 IU) , and alpha-lipoic acid (600 mg). all BID
  Vitamin E, 600IU: Vitamin C (1000 mg) , Vitamin E (600 IU) , and alpha-lipoic acid (600 mg). all BID
  Alpha Lipoic Acid, 600mg: Vitamin C (1000 mg) , Vitamin E (600 IU) , and alpha-lipoic acid (600 mg). all BID
- Protocol 2: BH4 (5mg): measurements at baseline and 3 hours following the single dose of 5mg/kg Kuvan® or sapropterin dihydrochloride which is a synthetic preparation of the dihydrochloride salt of naturally occurring tetrahydrobiopterin (BH4).BH4 has been shown in past studies to increase NO bioavailability.
  BH4: Kuvan® or sapropterin dihydrochloride is a synthetic preparation of the dihydrochloride salt of naturally occurring tetrahydrobiopterin (BH4). Subjects will receive an oral dose of 20 mg/kg of Kuvan® (Biomarin Pharmaceuticals Inc.)
- Protocol 2: BH4 (20mg): measurements at baseline and 3 hours following the single dose of 20mg/kg Kuvan® or sapropterin dihydrochloride which is a synthetic preparation of the dihydrochloride salt of naturally occurring tetrahydrobiopterin (BH4).BH4 has been shown in past studies to increase NO bioavailability.
  BH4: Kuvan® or sapropterin dihydrochloride is a synthetic preparation of the dihydrochloride salt of naturally occurring tetrahydrobiopterin (BH4). Subjects will receive an oral dose of 20 mg/kg of Kuvan® (Biomarin Pharmaceuticals Inc.)
- Healthy Controls: measurements were done with no intervention
Period: Overall Study
Arm/Group | Protocol 1: AOC | Protocol 2: BH4 (5mg) | Protocol 2: BH4 (20mg) | Healthy Controls
Started | 18 | 17 | 12 | 17
Completed | 18 | 17 | 12 | 17
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Protocol 1: AOC | Protocol 2: BH4 (5mg) | Protocol 2: BH4 (20mg) | Healthy Controls | Total
Number analyzed (Participants) | 18 | 17 | 12 | 17 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.9 (7.5) | 17 (7) | 19 (8) | 15.7 (5.2) | 17.3 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 6 | 9 | 35
  Male | 8 | 7 | 6 | 8 | 29
Height [Mean (Standard Deviation); unit: cm] | 158.6 (14.2) | 158.1 (14.1) | 162.1 (11.1) | 162.9 (14.7) | 160.3 (14.0)
Weight [Mean (Standard Deviation); unit: kg] | 53.1 (14.7) | 53.0 (14.6) | 57.8 (14.7) | 52.5 (16.5) | 53.8 (15.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Flow-Mediated Dilation (FMD)
Description: Brachial artery FMD induced by reactive hyperemia assessed vascular endothelial function at baseline and several hours after treatment.
Time Frame: pre-treatment Baseline and 2-3 hours post-treatment
Population: Participants included patients diagnosed with cystic fibrosis and healthy age-matched controls.
Measure: Mean (Standard Deviation); unit: percentage of change in FMD
Arm/Group | Protocol 1: AOC | Protocol 2: BH4 (5mg) | Protocol 2: BH4 (20mg) | Healthy Controls
Number analyzed (Participants) | 18 | 17 | 12 | 17
percentage of change in FMD
  Pre treatment | 5.64 (2.80) | 5.32 (3.53) | 6.29 (3.21) | 7.21 (3.17)
  Post treatment: number analyzed (Participants) | 18 | 17 | 12 | 0
  Post treatment | 7.58 (4.16) | 4.81 (2.83) | 7.39 (3.41) |

ADVERSE EVENTS:
Groups:
- Antioxidant Cocktail: CF Patients: measurements at baseline and 2 hours following the antioxidant cocktail that is comprised of over the counter vitamins (vitamin C 1000mg, vitamin E 600 IU, and alpha lipoic acid 600 mg) that will be given in two doses, 30 minutes apart.
  Vitamin C, 1000mg: Vitamin C (1000 mg) , Vitamin E (600 IU) , and alpha-lipoic acid (600 mg). all BID
  Vitamin E, 600IU: Vitamin C (1000 mg) , Vitamin E (600 IU) , and alpha-lipoic acid (600 mg). all BID
  Alpha Lipoic Acid, 600mg: Vitamin C (1000 mg) , Vitamin E (600 IU) , and alpha-lipoic acid (600 mg). all BID
- Antioxidant Cocktail: Healthy Controls: measurements at baseline and 2 hours following the antioxidant cocktail that is comprised of over the counter vitamins (vitamin C 1000mg, vitamin E 600 IU, and alpha lipoic acid 600 mg) that will be given in two doses, 30 minutes apart.
  Vitamin C, 1000mg: Vitamin C (1000 mg) , Vitamin E (600 IU) , and alpha-lipoic acid (600 mg). all BID
- Tetrahydrobiopterin (BH4): 5mg: measurements at baseline and 3 hours following the single dose of 5mg/kg Kuvan® or sapropterin dihydrochloride which is a synthetic preparation of the dihydrochloride salt of naturally occurring tetrahydrobiopterin (BH4).BH4 has been shown in past studies to increase NO bioavailability.
  BH4: Kuvan® or sapropterin dihydrochloride is a synthetic preparation of the dihydrochloride salt of naturally occurring tetrahydrobiopterin (BH4). Subjects will receive an oral dose of 20 mg/kg of Kuvan® (Biomarin Pharmaceuticals Inc.)
- Tetrahydrobiopterin (BH4): 20mg: measurements at baseline and 3 hours following the single dose of 20mg/kg Kuvan® or sapropterin dihydrochloride which is a synthetic preparation of the dihydrochloride salt of naturally occurring tetrahydrobiopterin (BH4).BH4 has been shown in past studies to increase NO bioavailability.
  BH4: Kuvan® or sapropterin dihydrochloride is a synthetic preparation of the dihydrochloride salt of naturally occurring tetrahydrobiopterin (BH4). Subjects will receive an oral dose of 20 mg/kg of Kuvan® (Biomarin Pharmaceuticals Inc.)
Arm/Group | Antioxidant Cocktail: CF Patients | Antioxidant Cocktail: Healthy Controls | Tetrahydrobiopterin (BH4): 5mg | Tetrahydrobiopterin (BH4): 20mg
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/17 | 0/12
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/17 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No